CLINICAL TRIAL: NCT02774590
Title: Timolol for the Treatment of Acne and Rosacea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00074049
Record Dates: First submitted 2016-05-09; First posted 2016-05-17 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-01

CONDITIONS: Acne Vulgaris; Rosacea
Keywords: Acne vulgaris; Rosacea
MeSH Terms: conditions — Acne Vulgaris; Rosacea | interventions — Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Timolol to split face for 8 weeks (Experimental): All 24 subjects will receive study drug and everyone will be randomized to which side of the face is treated with study drug first (right half-face versus left half-face). After 8 weeks of split-face treatment every night before bed, the subjects will be instructed to start treating both sides for another 8 weeks. Up to 30 subjects may be enrolled to ensure a target sample size of 24 (12 acne cases, 12 rosacea cases). This is an exploratory study. No part of this protocol will be considered routine care.
  Interventions: Drug: Timolol

INTERVENTIONS:
Drug: Timolol — Apply timolol on half of the participant's face for 8 weeks. Then treat both sides of face for 8 weeks.

SUMMARY:
This research is being done to determine the safety and tolerability of timolol in the treatment of acne and rosacea. The investigators will also look for specific biomolecular changes in acne or rosacea skin when it is exposed to timolol.

Timolol is approved by the Food and Drug Administration (FDA) for the treatment of glaucoma. In dermatology, it has been used as a treatment to decrease the size of vascular (blood vessel) malformations in infant skin. Timolol is not approved for use in acne or rosacea and its use in this study is investigational.

Many people with rosacea have telangiectasias which are small, red dilated blood vessels on the skin. They also suffer from flushing and acne-like lesions. Better treatments than those currently available are desired.

Acne vulgaris, or acne, is another chronic inflammatory and very common skin disease that affects about 8 out of 10 young adults and adolescents. Signs of acne include papules and blackheads that are often called primary lesions because they represent an active form of the disease. There are also secondary lesions that can form later; they are known as acne scars

DETAILED DESCRIPTION:
Rosacea affects roughly 16 million Americans who desire better treatments than those currently available. Acne vulgaris, another chronic inflammatory skin disorder, mainly affects teenagers but also affects 20-40% of adults. Investigating potential new treatments will not only satisfy a clinical need, but also offers the opportunity to learn about the pathogenesis of the disease and skin biology. The purpose of this study is to investigate the possible role of timolol as a therapy for the erythema and papules associated with acne and rosacea. It has been shown that timolol is beneficial and safe to treat infantile hemangiomas. The investigators hypothesize that it may also be safe and effective in the treatment of acne and rosacea.

In a single experiment where the test case was the PI (a practicing physician), the investigators treated his rosacea with timolol for this off-label indication and have noticed an improvement in flushing and an unexpected improvement in acneiform eruptions associated with the rosacea. After 30 days, less flushing and acneiform lesions were noted on the treated right side compared to the left side . Similarly, at 60 days after treatment, as visualized by infrared imaging, significantly less inflammation and flushing was noted on the treated right side even outside of episodes of flushing. The improvement was durable, such that after a 60 day washout, improvements were still noted. In summary, during testing of the PI as a case subject, timolol appeared effective, safe, and with some disease-remissive effects.

Our aim is to conduct a 16 week split-face pilot study with up to 30 patients who have a diagnosis of either inflammatory acne or rosacea to assess whether timolol maleate effectively reduces erythema, flushing, telangiectasias, and/or papules. The investigators also propose to biopsy a subset of our study patients to examine the biological activity in the skin before and after treatment. The investigators are particularly interested in studying epigenetic DNA methylation abnormalities in these conditions at baseline to compare to normal subjects and as a result of therapy.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, must be medically able to undergo the administration of study material
* Be able to comprehend the informed consent document and provide consent for participation
* Females of childbearing potential must:

  * Not be pregnant by subjective report
  * agree to not become pregnant or breastfeed for the period of the study through 1 month after completion of the study
  * be willing to use a reliable form of contraception during the study
* Be willing and able to comply with the scheduled visits and other study procedures for the duration of the study.
* Be willing not to take any other medicine for acne or rosacea during the study
* Acne specific inclusion criteria:

  o 10-100 noninflammatory, 20-50 inflammatory lesions (nose excluded)
* Rosacea specific inclusion criteria:

  * History of frequent flushing
  * Skin erythema - Positive (not negative) chromometer minimum reading difference when subtracting nonaffected reading from affected reading.

Goal would be greater than 1 unit difference between red areas. For example, the red area (average 17.7 Chroma Meter a) and nonaffected areas (average 14.1 Chroma Meter a), yields in an optimum scenario greater than 3 point difference in this example (in subjects with average Chromometer L value averaging 56.6-59.6). Example from (Helfrich et al., 2015).

o Presence of inflammatory papules

Exclusion Criteria:

* Having received any investigational drug within 30 days prior to study entry
* An allergy history to any study materials including any beta-blockers.
* Pregnant, lactating, or trying to become pregnant
* Severe depression
* Hypotension or history
* Bradycardia or history
* History of Cardiac Heart Failure
* History of Myocardial infarction
* History of heart arrhythmia
* Asthma or Bronchospasm or history
* Rosacea specific exclusion criteria:

Recent topicals within 3 weeks Oral rosacea medications such as antibiotics within 3 weeks • Acne specific exclusion criteria: nodular acne man with beard which interferes with clinical evaluation history of Accutane Oral contraceptive pills changes last 3 months Topical retinoid within 4 weeks Cosmetic procedures (like facial or peels) for 4 weeks Photodynamic therapy , laser therapy or microdermabrasion for 4 weeks Other topicals or oral acne medications such as antibiotics within 3 weeks

o Biopsy volunteer specific exclusion criteria: History of keloids History of hypertrophic scars Allergy to lidocaine or epinephrine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of timolol for acne and rosacea as assessed by subject report | 8 weeks
  To determine the safety and tolerability of Timolol in the treatment of acne and rosacea
Safety and tolerability of timolol for acne and rosacea as assessed by physician assessment | 8 weeks
  To determine the safety and tolerability of Timolol in the treatment of acne and rosacea

SECONDARY OUTCOMES:
Decrease of rosacea activity as assessed through visual assessments (photographs, chronometer, patient report and physician examination) | 8 weeks
  In rosacea, to measure decreases of disease activity-- redness.
Decrease of acne activity: papules | 8 weeks
  In acne, to measure decreases of disease activity: papules
Test if the DNA methylation patterns are corrected following clinical improvement as assessed by microarray | 8 weeks
  In both conditions, test if the DNA methylation patterns specific to each is corrected following clinical improvement after timolol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Garza, MD, PhD, Principal Investigator — Johns Hopkins Dermatology
Locations (1):
- Johns Hopkins Dermatology Department, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Following publication the investigators will honor all requests for original data

REFERENCES:
- [Result] Tsai J, Chien AL, Kim N, Rachidi S, Connolly BM, Lim H, Alessi Cesar SS, Kang S, Garza LA. Topical timolol 0.5% gel-forming solution for erythema in rosacea: A quantitative, split-face, randomized, and rater-masked pilot clinical trial. J Am Acad Dermatol. 2021 Oct;85(4):1044-1046. doi: 10.1016/j.jaad.2021.01.098. Epub 2021 Feb 3. No abstract available. PMID 33548303